CLINICAL TRIAL: NCT01323569
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Abuse Potential of Sativex in Subjects With a History of Recreational Marijuana Use
Brief Title: Abuse Potential of Sativex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GWCP0605
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Evaluation of Abuse Potential of Sativex
Keywords: Sativex; Cannabinoids; Abuse potential; Addiction
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sativex 4 sprays (Experimental)
  Interventions: Drug: Sativex
- Sativex 8 sprays (Experimental)
  Interventions: Drug: Sativex
- Sativex 16 sprays (Experimental)
  Interventions: Drug: Sativex
- Marinol low dose (Active Comparator)
  Interventions: Drug: Marinol
- Marinol high dose (Active Comparator)
  Interventions: Drug: Marinol

INTERVENTIONS:
Drug: Sativex — Sativex dose level 1: 10.8 mg THC/10 mg CBD (4 sprays) + 12 placebo sprays + 4 placebo capsules.
  Arms: Sativex 4 sprays
Drug: Sativex — Sativex dose level 2: 21.6 mg THC/20 mg CBD (8 sprays) + 8 placebo sprays + 4 placebo capsules
  Arms: Sativex 8 sprays
Drug: Sativex — Sativex dose level 3: 43.2 mg THC/40 mg CBD (16 sprays) + 4 placebo capsules
  Arms: Sativex 16 sprays
Drug: Placebo — 16 placebo sprays and 4 placebo capsules
  Arms: Placebo
Drug: Marinol — Marinol dose level 1: 20 mg THC (2 marinol capsules) + 2 placebo capsules + 16 placebo sprays
  Arms: Marinol low dose
Drug: Marinol — Marinol dose level 2: 40 mg THC (4 marinol capsules) + 16 placebo sprays
  Arms: Marinol high dose

SUMMARY:
This crossover study with six treatment sessions is to evaluate the abuse potential of three doses of Sativex as compared to Marinol and placebo, in subjects with a history of recreational marijuana use.

DETAILED DESCRIPTION:
Subjects attended a two-session, randomized, double-blind, crossover qualification in which they received the positive control drug (Marinol 30 mg) and matching placebo 48 hours apart in a randomized fashion. To qualify, subjects must have discriminated between Marinol and placebo.

Eligible subjects then went on to the main study divided into six treatment sessions each separated by 7-21 days.

Serial pharmacodynamic evaluations were taken at each treatment session as well as occasional pharmacokinetic blood samples to verify proof of exposure. In addition, safety monitoring included regular assessments of vital signs, telemetry, 12-lead ECG, clinical laboratory tests and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 19 to 45 years of age, inclusive.
* Current recreational marijuana users, defined as the use of smoked marijuana, hashish, or oral THC, at least once a week for the 3 months prior to screening and, on at least one occasion, four times in a given week in the 3 months prior to screening.
* Body mass index within the range of 19 to 30 kg/m2 inclusive and a minimum weight of at least 50 kg at screening.
* Free of any clinically significant abnormality, assessed at screening, on the basis of medical history, vital signs, physical examination, 12-lead ECG, and clinical laboratory tests, including haematology, clinical chemistry, urinalysis, and serology, as judged by the investigator or designee.
* A positive urine THC drug screen at screening and qualification, which was confirmed by quantitative analysis; the level must have been at least 50 ng of THC/mL.
* A negative urine drug screen for cocaine, opiates, amphetamine, and benzodiazepines upon admission to the screening, qualification session, or treatment sessions. Subjects who had a positive urine drug screen upon presentation to a study visit could have been rescheduled for another session at the discretion of the investigator.
* All female subjects were required to have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the qualification session and to each drug treatment session.
* Subjects with reproductive potential could be entered into the study if they had been using and were willing to continue to use two methods of contraception for the duration of the study. These methods included male condom for men in addition to an oral contraceptive, contraceptive implant or injection, intrauterine device, diaphragm, or a contraceptive sponge for women. Adequate protection, as defined above, had to have been used for at least 1 month prior to screening for all, with the exception of oral contraceptives, which should have been used for at least 3 months prior to screening. These methods had to be continually used for 30 days after the end of the study. Subjects that had been surgically sterilized (tubal ligation, hysterectomy, or vasectomy) or had been post-menopausal for at least 2 years (by history) were not considered to be of reproductive potential.
* Subjects had to pass a qualification session.
* Must have understood and provided written informed consent, prior to initiation of any protocol-specific procedures.
* Subjects were able to comply with study procedures.
* Negative breath alcohol test. Subjects who had a positive breath alcohol test could have been rescheduled at the discretion of the investigator.

Exclusion Criteria:

* History or presence of drug or alcohol dependence (excluding nicotine and caffeine), including subjects who had ever been in a drug rehabilitation program.
* Clinically important impairment or dysfunction of any body system, including, but not limited to, the following: cardiovascular, haematological, hepatic, gastrointestinal, renal, pulmonary, or neurological, as judged by the investigator or designee.
* Any known or suspected history (including family history) of schizophrenia or other psychotic illness. Presence or history of a psychiatric disorder, organic brain disorder, or seizure disorder that was deemed clinically significant by the investigator.
* History of hypersensitivity or allergy to cannabinoids, cannabis and/or its metabolites, to the study drug excipients, or to similar compounds (propylene glycol, ethanol, peppermint, and sesame oils) or allergic reactions to any other medication.
* Consumed caffeine-containing beverages in excess of 450 mg of caffeine (e.g. 5 cups of tea or 3 cups of regular coffee or 8 cans of cola) per day in the 6 months prior to screening.
* Consumed greater than 20 cigarettes per day.
* Treatment with another investigational or non-approved drug, within 4 weeks prior to the start of qualification session dosing (Day 1).
* Donated or lost blood (>100 mL) within the 30 days prior to screening.
* Female subjects who were pregnant or lactating or who were planning to become pregnant within 60 days of last study drug administration.
* Used prescription drugs (except oral contraceptives or sex hormone replacement), including smoked THC for medicinal purposes, within 14 days of the qualification session and for the duration of the study, unless in the opinion of the investigator (or designee), the medication received would not interfere with the study procedures or data integrity or compromise the safety of the subject.
* Used non-prescription drugs or natural health products other than acetaminophen up to 2 g per day or vitamin or mineral supplements (including mega dose vitamin therapy), within 7 days prior to the qualification session, and for the duration of the study, unless in the opinion of the investigator (or designee), the medication received would not interfere with the study procedures or data integrity or compromise the safety of the subject.
* Uncontrolled hypertension at screening that was judged as clinically significant by the investigator (or designee).
* Subjects who, in the opinion of the investigator (or designee). were not willing, able or capable of following the study schedule for any reason.
* Subjects who were positive for or were being treated for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Subjects facing current or pending legal charges.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Comparison of Subjective Drug Value (SDV)(Balance of effects) between Marinol and Sativex | Recorded at 6, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg.
Comparison of Bipolar Drug Liking VAS (Balance of effects) between Marinol and Sativex | Recorded at 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg.
Comparison of Addiction Research Centre Inventory (ARCI) MBG (Positive effects) between Marinol and Sativex | Recorded at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg.

SECONDARY OUTCOMES:
Comparison of Balance of Effects VASs between Marinol and Sativex | Recorded at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg. for each of Overall Drug Liking VAS, Take Drug Again VAS, Pleasant Mental state VAS, and Pleasant Physical state VAS.
Comparison of Positive Effects VASs between Marinol and Sativex | Recorded at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg; for each of Good effects VAS and High VAS.
Comparison of Cannabinoid Effects between Marinol and Sativex | Recorded at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg; for each of ARCI Marijuana, Stoned VAS, Mellow VAS, Clarity VAS, and Hungry VAS.
Comparison of Negative Effects Scores between Marinol and Sativex | Recordedat 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg; for each of ARCI Lysergic Acid Diethylamide, Bad Effects VAS, Nausea VAS, Feeling Sick VAS, and Room Spinning VAS.
Comparison of Other Effects Scores between Marinol and Sativex | Recorded pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study arm
  Mean difference in Mean peak effect (Emax) between:
  Marinol 20 mg vs Sativex 21.6 mg; Marinol 20 mg vs Sativex 43.2 mg; Marinol 40 mg vs Sativex 43.2 mg; for each of: Any effects VAS, Dizziness VAS, ARCI Pentobarbital-Chlorpromazine-Alcohol Group, Drowsiness VAS, ARCI Benzedrine Group, and ARCI Amphetamine, Drug similarity VASs, Choice Reaction Time, Divided Attention, Sternberg short-term memory tests.
Area under the concentration-time curve from 0 to 8.5 hours post-dose for plasma THC, CBD, and 11-hydroxy-THC. | Pre-dose and at 1, 4, and 8 hours during each study visit
Adverse Events | Recorded pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours during each study visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- DecisionLine Clinical Research Corporation, Toronto, Ontario, Canada

REFERENCES:
- [Result] Schoedel KA, Chen N, Hilliard A, White L, Stott C, Russo E, Wright S, Guy G, Romach MK, Sellers EM. A randomized, double-blind, placebo-controlled, crossover study to evaluate the subjective abuse potential and cognitive effects of nabiximols oromucosal spray in subjects with a history of recreational cannabis use. Hum Psychopharmacol. 2011 Apr;26(3):224-36. doi: 10.1002/hup.1196. PMID 21671456